CLINICAL TRIAL: NCT02242019
Title: An Evaluation of the Effect of the Erchonia LUNULA on Treating Toenail Onychomycosis
Brief Title: Study of Erchonia Low Level Laser Light Therapy to Treat Toenail Fungus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_TFRS_004
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erchonia LUNULA (Experimental): The Erchonia LUNULA emits both red light (635 nm) and blue light (405 nm) to the affected toenail for 12 minutes per treatment for 4 treatments, each treatment one week apart.
  Interventions: Device: Erchonia LUNULA

INTERVENTIONS:
Device: Erchonia LUNULA — The Erchonia LUNULA is administered to the infected toes for 12 minutes per treatment for 4 treatments, each treatment one week apart.

SUMMARY:
The purpose of this study is to determine whether low level laser light therapy is effective in the treatment of toenail onychomycosis.

DETAILED DESCRIPTION:
An infection of toenail fungus, or onychomycosis, typically occurs when fungi (most commonly dermatophytes) infect the nail, but may also be caused by yeasts and molds. The nail fungal infection usually begins as a white or yellow spot under the tip of the toenail and then spreads deeper into the nail causing discoloration, thickening and the development of crumbling edges to the nail which can be unsightly and painful and may produce serious physical and occupational limitations. Onychomycosis can also have a detrimental effect on an individual's quality of life, affecting their psychosocial and emotional wellbeing.

Onychomycosis can be difficult to treat, and infections recur easily. Toenail fungus affects approximately 23 million adults (about 10%) in the United States. It is more common among older adults and tends to affect men more than women. Potential complications of onychomycosis include pain, permanent damage to the nails and serious infections that can spread beyond the feet.

Currently available treatments for onychomycosis include oral antifungal medications (Lamisil, Sporanox); antifungal nail polish (Penlac); topical over-the-counter antifungal creams; photodynamic therapy and in more severe cases, surgery to remove the nail. However, there is no perfect cure for toenail fungus. Even the most effective oral medications are only successful about half of the time, and topical medications are successful less than 10% of the time. In addition, clearance of the infection and growth of new clear nail can be slow, and the rate of recurrence of infection is high. Antifungal drugs may also cause side effects ranging from skin rashes to liver damage.

Therefore, the need for a more effective and lasting cure is evident. Recently, research has found laser therapy to show promise as a novel alternative treatment for toenail onychomycosis. Unlike medication-driven treatments, laser therapy presents minimal risk of side effects. Laser therapy is applied to toenail onychomycosis by shining a laser light through the toenail. The laser light vaporizes the fungus while leaving the skin and surrounding tissue unharmed.

Low level laser light therapy operates under the principle of photochemistry with a photoacceptor molecule absorbing the emitted photons and inducing a biological cascade. Like our eukaryotic cell, fungi contain the highly complex organelle the mitochondria, which is responsible for the manufacturing of the energy molecule Adenosine triphosphate (ATP). Within the inner mitochondrial membrane is cytochrome c oxidase, an identified photoacceptor molecule. It is believed that laser therapy could perhaps provide a means to photo-destroy the fungi responsible for onychomycosis by inducing the release of highly reactive superoxides. Moreover, laser therapy has been shown to promote superoxide dismutase (SOD), a process responsible for the destruction of foreign invaders. Extracellular release of low levels of mediators associated with SOD can increase the expression of chemokines, cytokines, and endothelial leukocyte adhesion molecules, amplifying the cascade that elicits the inflammatory response. The physiologic function of hydrogen peroxide, superoxide anion, and hydroxyl free radical is to destroy phagocytosed microbes. By enhancing the natural processes of the immune system and impacting the structural integrity of the fungi strain, it is believed that laser therapy may provide a means for clinicians to effectively treat onychomycosis without the onset of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Onychomycosis present in at least one great toenail, identified as current bacterial/fungal infection classified by the investigator as onychomycosis, with the nail presenting positive on visual inspection for somewhat thickened nail plate with a cloudy appearance and some discoloration (white to yellow to brown).
* Subject is willing and able to refrain from employing other (non-study) treatments (traditional or alternative) for his or her toenail onychomycosis throughout study participation.
* Subject is willing and able to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers throughout study participation.

Exclusion Criteria:

* Spikes of disease extending to nail matrix in the affected great toenail(s).
* Infection involving lunula of the affected toenail(s), e.g., genetic nail disorders, primentary disorders.
* Affected great toenail(s) has less than 2mm clear (unaffected) nail plate length beyond the proximal fold.
* Presence of dermatophytoma (defined as thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the affected great toenail(s).
* Chronic plantar (moccasin) tinea pedis.
* History of current or past psoriasis of the skin and/or nails.
* Concurrent lichen planus.
* Onychogryphosis.
* Any of the following conditions of the affected great toenail(s) is present: proximal subungual onychomycosis; white superficial onychomycosis; dermatophytoma or "yellow spike/streak"; exclusively lateral disease
* Confounding problems/abnormalities of the great toenail(s).
* Any abnormality of the affected great toenail(s) that could prevent a normal appearing nail if clearing of infection is achieved.
* Inability for the affected great toenail(s) to become normal in the opinion of the investigator.
* History of multiple repeated failures with previous therapies for onychomycosis.
* Trauma to the affected great toenail(s).
* Use of oral antifungal agents in the past 6 months.
* Use of topical antifungal agents in the past 1 month.
* Prior surgical treatment of the affected great toe(s).
* Subject is unwilling or unable to refrain from employing other (non-study) treatments (traditional and alternative) for his or her toenail onychomycosis throughout study participation.
* Subject is unwilling or unable to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers until the end of study participation.
* Cancer and/or treatment of any type of cancer within the last six months.
* Peripheral vascular disease or peripheral circulatory impairment.
* History of uncontrolled diabetes mellitus.
* Known immunodeficiency.
* Known sensitivity, or contraindication, to light therapy.
* Pregnant, breast feeding, or planning pregnancy prior to the end of study participation.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirements and/or record the necessary study measurements.
* Involvement in litigation and/or receiving disability benefits related in any way to the parameters of the study.
* Participation in a clinical study or other type of research in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sullivan, Podiatry, Principal Investigator
Locations (1):
- Midleton Foot Clinical, Midleton, Co. Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia LUNULA
Started | 109
Completed | 109
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia LUNULA
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.89 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 109
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 109
Duration of toenail onychomycosis Involvement [Mean (Standard Deviation); unit: months] | 25.99 (18.43)
Percent Toenail Onychomycosis Disease Involvement [Mean (Standard Deviation); unit: percentage of toenail] | 63.21 (23.88)
Millimeter (mm) of Clear Nail From the Lunula [Mean (Standard Deviation); unit: millimeters (mm)] | 5.90 (4.58)

OUTCOME MEASURES:

1. Primary Outcome: Number of Toenails Attaining 3 Millimeters (mm) or More of Clear Nail Growth
Description: Individual toenail success criteria was defined as 3 millimeter (mm) or more of clear nail growth at 36 weeks post-procedure administration as evaluated relative to baseline. Overall study success criteria was defined as an 60% or more of treated toenails meeting the individual success criteria.
Time Frame: Baseline and 36 Weeks
Measure: Number; unit: toenails
Units Other Than Participants: toenails
Arm/Group | Erchonia LUNULA
Number analyzed (Participants) | 109
Number analyzed (toenails) | 139
toenails | 134

2. Secondary Outcome: Change in Percent (%) of Onychomycosis Disease Involvement
Description: The percent (%) of the toenail that had onychomycosis disease involvement was determined. Change in the % of toenail onychomycosis disease involvement was calculated as the difference in the % of toenail onychomycosis disease involvement from baseline measurement to the measurement at 36 weeks after the end of the procedure administration phase. A decrease in the % of toenail onychomycosis disease involvement between the two measurement points indicates that the toenail onychomycosis involvement has decreased and is positive for study success. An increase in the % of toenail onychomycosis disease involvement between the two measurement points indicates that the toenail onychomycosis involvement has increased and is negative for study success.
Time Frame: Baseline and 36 Weeks
Measure: Mean (Standard Deviation); unit: percentage of disease involvement
Units Other Than Participants: toenails
Arm/Group | Erchonia LUNULA
Number analyzed (Participants) | 109
Number analyzed (toenails) | 139
percentage of disease involvement | 57.76 (21.97)
Statistical Analysis 1: Comparison: Erchonia LUNULA; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Primary Outcome: Change in Millimeters (mm) of Clear Nail Bed
Description: Millimeter (mm) of clear nail from the base of the toenail was determined from digital photographs of the toenail using a computer program. Change in mm of clear nail bed was calculated as the difference in mm of clear nail bed from baseline measurement to the measurement at 36 weeks after the end of the procedure administration phase. An increase in mm of clear nail between the two measurement points indicates that the toenail has improved and is positive for study success. A decrease in mm of clear nail between the two measurement points indicates that the toenail has worsened and is negative for study success.
Time Frame: Baseline and 36 Weeks
Population: Some subjects had multiple toenails with onychomycosis disease involvement that were treated and analyzed, resulting in a total of 139 study toenails being analyzed.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: toenails
Arm/Group | Erchonia LUNULA
Number analyzed (Participants) | 109
Number analyzed (toenails) | 139
millimeters (mm) | 8.36 (4.08)
Statistical Analysis 1: Comparison: Erchonia LUNULA; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Erchonia LUNULA
Serious Adverse Events (participants affected / at risk) | 0/109
Other Adverse Events (participants affected / at risk) | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No